CLINICAL TRIAL: NCT00268060
Title: Baby R. Case Report Proposal
Brief Title: Infant Medical Records: Case Report Proposal
Status: Terminated | Type: Observational
Sponsor: Children's Healthcare of Atlanta (Other)
Other Study IDs: 05-050
Record Dates: First submitted 2005-12-20; First posted 2005-12-22 (Estimated); Last update posted 2007-05-07 (Estimated); Status verified 2007-05

CONDITIONS: Congenital Disorders
Keywords: pediatric; cardiac; Long QT Syndrome; Pacemaker; Herg mutation
MeSH Terms: conditions — Congenital, Hereditary, and Neonatal Diseases and Abnormalities; Long QT Syndrome

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Retrospective

SUMMARY:
Infants with congenital long QT syndrome (LQTS) and 2:1 atrioventricular block (AVB) have been recognized as a clinical subset of children with LQTS.

The purpose of this study is to describe the clinical course and outcome of a patient with congenital long QT syndrome (LQTS).

DETAILED DESCRIPTION:
It has been previously reported that 2:1 AVB in neonatal LQTS seems preferentially associated with HERG mutations . It has also been reported in association with the SCN5A gene. We report on a neonate with congenital LQTS and congenital complete heart block who experienced frequent episodes of torades des pointe and ventricular tachycardia, which, over the first 2 days of life, was recalcitrant to traditional therapy of beta-blockers and other antiarrhythmics. Eventually hypotension necessitated the use of an epinephrine infusion, which halted the ventricular tachyarrhythmias. A pacemaker was implanted once the infant was stable and, currently, he is thriving. Genetic analysis revealed a HERG mutation.

For this study, we will need access to the infant's inpatient and outpatient medical records at Children's Healthcare of Atlanta at Egleston Children's Hospital and Sibley Heart Center Cardiology to include his age, date of birth, medical record number, inpatient labs, inpatient echo reports, outpatient echo reports, inpatient and outpatient EKG's, inpatient pharmacy records, the results of his genetic analysis, his history and physical, transfer notes, daily progress notes, consultation reports and operative reports from his admission beginning 9/30/04.

ELIGIBILITY:
Inclusion Criteria:

* Congenital long QT Syndrome single case report

Exclusion Criteria:

* Single case report

Max Age: 21 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1
Dates: Start 2004-09

CONTACTS AND LOCATIONS:
Overall Officials: Tracy Froehlich, MD, Principal Investigator — Children's Healthcare of Atlanta
Locations (1):
- Chldren's Healthcare of Atlanta, Atlanta, Georgia, United States